CLINICAL TRIAL: NCT03276364
Title: The Impact of Point-of-Care Ultrasound Performed by Trainees to Improve the Prediction of Fluid Responsiveness in Patients With Shock
Brief Title: The Impact of Point-of-Care Ultrasound
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: Beth Israel Medical Center (Other)
Responsible Party: Principal Investigator, Daniel G. Fein, Assistant Professor of Medicine, Montefiore Medical Center
Other Study IDs: 206-13
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Ultrasound; Shock
MeSH Terms: conditions — Shock | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Shock
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Point-of-care ultrasound examination by pulmonary and critical care fellow

SUMMARY:
Point-of-care ultrasound (POCUS) has been found to be useful for aiding in the prediction of fluid responsiveness. It is unknown if trainees can effectively utilize this tool to improve their assessment of fluid responsiveness.

In this prospective, observational study, pulmonary and critical care fellows are asked to make 2 assessments of fluid responsiveness in adults with shock: (1) based on clinical exam alone (Clinical) and (2) after performing a POCUS (Clinical + US). The accuracy of their pre- and post-ultrasound assessments are compared using a bioreactance monitor and passive leg raise test as the gold standard of fluid responsiveness in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 or older admitted to the MICU with a diagnosis of shock while a fellow was on duty.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Could undergo both a POCUS and bioreactance assessment within 6 hours of admission from the emergency department or transfer from a medical floor.
  * Shock was defined as either systolic blood pressure less than 90 mmHg or 40 mmHg below baseline, necessity for vasopressors to maintain mean arterial pressure greater than 65 mmHg, or any evidence of acute organ hypoperfusion that was evident at the time of study enrollment as judged by the treating physician.
  * The patient needed to be in shock at the time of POCUS and bioreactance testing at time of enrollment in order to be included.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2014-07-21 (Actual); Primary Completion 2015-04-17 (Actual); Study Completion 2015-04-17 (Actual)

PRIMARY OUTCOMES:
Fluid responsiveness | Immediately subsequent to performance of a point-of-care ultrasound exam
  Increase of stroke volume index greater than 10% following passive leg raise testing

IPD SHARING:
Plan to Share IPD: Undecided